CLINICAL TRIAL: NCT07282548
Title: A Prospective Real-World Study Evaluating Objective Response Rate and Duration of Response of Tazemetostat Monotherapy in Patients With Relapsed or Refractory Follicular Lymphoma Following at Least Two Prior Lines of Treatment
Brief Title: Study of Tazemetostat in Adults With Follicular Lymphoma Previously Treated With at Least Two Therapies
Status: Not yet recruiting | Type: Observational
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Other Study IDs: CLIN-60200-456
Record Dates: First submitted 2025-11-27; First posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Tazemetostat Monotherapy Group: Participants with relapsed or refractory follicular lymphoma (grades 1, 2, or 3A) who have received at least two prior lines of systemic therapy and are prescribed tazemetostat monotherapy in accordance with the approved U.S. Prescribing Information. Tazemetostat is administered orally at 800 mg twice daily, as per routine clinical practice. Treatment continues until disease progression, unacceptable toxicity, or other discontinuation criteria are met.

SUMMARY:
This study aims to evaluate how well the effectiveness of the medicine Tazemetostat works in adults with relapsed/refractory follicular lymphoma, a slow-growing type of blood cancer that affects a kind of white blood cell called lymphocytes.

All participants will receive Tazemetostat as prescribed by their doctor in the routine clinical practice.

The study will observe how participants respond to the treatment, how long the response lasts, and monitor safety, side effects and how well participants tolerate the treatment.

DETAILED DESCRIPTION:
The results will be analyzed based on whether or not participants have a mutation in the Enhancer of zeste homolog 2 (EZH2) gene (known as EZH2 wild-type).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Histologically confirmed follicular lymphoma grades 1, 2, or 3A
* At least two prior lines of systemic therapy
* Prescribed tazemetostat according to United States prescribing information (USPI)
* Known or planned EZH2 mutation status
* Signed informed consent

Exclusion Criteria:

* Grade 3B or transformed follicular lymphoma
* Other hematologic malignancies
* Use of strong/moderate Cytochrome P450 (CYP3A) inhibitors
* Pregnant or breastfeeding
* Participation in another investigational program

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This study will enroll approximately 63 adult participants with relapsed or refractory follicular lymphoma (FL) grades 1, 2, or 3A. All participants must have received at least two prior lines of systemic therapy and be prescribed tazemetostat monotherapy in accordance with the approved U.S. Prescribing Information. The population includes both EZH2 wild-type and mutant cases, with mutation status either known at enrollment or determined during the study. Participants will be recruited from U.S.-based community oncology practices, hospital systems, and academic medical centers.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2031-06-30 (Estimated); Study Completion 2031-06-30 (Estimated)

PRIMARY OUTCOMES:
Real-world Objective Response Rate (rwORR) stratified by EZH2 mutation status. | Fom first dose to end of study participation, which may range from 1 day to up to 5 years.
  rwORR is defined as the percentage of participants with a best overall response of complete response (CR) or partial response (PR), assessed by the investigator using the Lugano 2014 classification.

SECONDARY OUTCOMES:
Real-world Best Overall Response (rwBOR) stratified by EZH2 mutation status. | From first dose to end of study participation, which may range from 1 day to up to 5 years.
  rwBOR is defined as the best response assessed by the investigator using Lugano 2014 classification recorded from the start of treatment until disease progression or recurrence
Real-world Duration of Response (rwDOR) stratified by EZH2 mutation status. | Fom first dose to end of study participation, which may range from 1 day to up to 5 years.
  rwDOR is defined as the time from the first documented evidence of CR or PR until disease progression or death from any cause.
Real-world Progression-Free Survival (rwPFS) stratified by EZH2 mutation status. | Fom first dose to end of study participation, which may range from 1 day to up to 5 years.
  rwPFS is defined as the time from the start of treatment to the date of first documented disease progression or death from any cause.
Real-world Disease Control Rate (rwDCR) stratified by EZH2 mutation status. | Fom first dose to end of study participation, which may range from 1 day to up to 5 years.
  rwDCR is defined as the percentage of participants with CR, PR, or stable disease (SD) as their best response.
Percentage of participants starting at each initial dose level stratified by EZH2 mutation status. | At Day 1
Percentage of participants with dose reductions and reasons for reduction stratified by EZH2 mutation status. | Fom first dose to end of study participation, which may range from 1 day to up to 5 years.
Duration of treatment (in days/months) stratified by EZH2 mutation status. | Fom first dose to end of study participation, which may range from 1 day to up to 5 years.
Percentage of participants with treatment interruptions and associated reasons stratified by EZH2 mutation status. | Fom first dose to end of study participation, which may range from 1 day to up to 5 years.
Percentage of participants with treatment discontinuation and associated reasons stratified by EZH2 mutation status. | Fom first dose to end of study participation, which may range from 1 day to up to 5 years.
Percentage of participants receiving subsequent systemic therapy after Tazemetostat stratified by EZH2 mutation status. | Fom last dose to end of study participation (up to 5 years).
Percentage of participants experiencing Treatment Emergent Adverse Events (TEAEs), including Adverse Drug Reactions (ADRs), Serious Adverse Events (SAEs), Adverse Events of Special Interest (AESIs) | From first dose until 30 days after last dose.
  An Adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. A TEAE is an AE for which the start date is on or after the date that the intervention began, or it was present prior to receiving the intervention but the intensity increased during the active phase of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications.
  Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the United States (US) and/or European Union (EU).
Access Criteria: Further details on Ipsen's sharing criteria and process for sharing are available here (https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/).
URL: https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/